CLINICAL TRIAL: NCT03811080
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-Group, Phase 3, Therapeutic Confirmatory Clinical Trial to Evaluate the Efficacy and Safety of DWP14012 in Patients With Non-Erosive Gastroesophageal Reflux Disease
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 in Patients With Non Erosive Reflux Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP14012302
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Non-Erosive Gastroesophageal Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWP14012 A mg (Experimental): DWP14012 A mg, tablet, once daily, oral administration for up to 4 weeks
  Interventions: Drug: DWP14012 A mg
- DWP14012 B mg (Experimental): DWP14012 B mg, tablet, once daily, oral administration for up to 4 weeks
  Interventions: Drug: DWP14012 B mg
- Placebo (Placebo Comparator): Placebo, tablet, once daily, oral administration for up to 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DWP14012 A mg — The participants will receive treatment of DWP14012 A mg, tablet, orally, once daily and DWP14012 B mg placebo-matching tablet, orally, once daily for up to 4 weeks.
  Arms: DWP14012 A mg
Drug: DWP14012 B mg — The participants will receive treatment of DWP14012 B mg, tablet, orally, once daily and DWP14012 A mg placebo-matching tablet, orally, once daily for up to 4 weeks.
  Arms: DWP14012 B mg
Drug: Placebo — The participants will receive treatment of DWP14012 A mg placebo-matching tablet, orally, once daily and DWP14012 B mg placebo-matching tablet, orally, once daily for up to 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the superiority of efficacy of DWP14012, once daily (QD), compared to placebo in patients with non-erosive reflux disease at Week 4.

DETAILED DESCRIPTION:
This is a multi-center, double blind, randomized, placebo-controlled, parallel-group, phase 3 study. Subjects will be randomly assigned to one of the three treatment groups (DWP14012 A mg or DWP14012 B mg or placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 20 and 75 years
2. Subjects who were not observed mucosal break according to the LA classification(LA grade) on the EGD
3. Subjects who had experienced major symptom within 3 months
4. Subjects who had experienced major symptom within 7 days before randomization. Entry into study also required that patients had experienced at least mild symptoms on at least 2 days/week or at least moderate symptoms on at least 1 day/week
5. Subjects who is able to understand and follow the instructions
6. Subjects who voluntarily signed written informed consent form

Exclusion Criteria:

1. Subjects who have Barrett's esophagus, gastroesophageal varices, esophageal stenosis, ulcer stenosis, active gastric ulcer, gastrointestinal bleeding or malignant tumor confirmed by endoscopy
2. Subjects who have erosive esophagitis, acute upper gastrointestinal bleeding, gastric ulcers or duodenal ulcers within 2 months before Visit 1
3. Subjects diagnosed with functional dyspepsia, primary esophageal motility disorder, IBS, IBD in the last 3 months
4. Subjects who have a history of gastric acid suppression surgery or gastroesophageal surgery
5. Subjects with Zollinger-Ellison syndrome
6. Subjects with eosinophilic esophagitis
7. Subjects with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease .

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
1. Percentage of patients with complete resolution of major symptoms (heartburn and acid regurgitation) at 4-week | 4 week
  defined as no episodes of symptom during the last 7 days of treatment, using Reflux Disease Questionnaire(RDQ)

SECONDARY OUTCOMES:
Reflux disease symptom assessment using RDQ(Reflux disease questionnaire) | 2 week, 4 week
Reflux disease symptom assessment using Subject diary | 4 week
Quality of Life assessment using PAGI-QoL | 4 week
Use of rescue medication | 4 week

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea